CLINICAL TRIAL: NCT03298880
Title: Testing of a Valsalva Assist Device (VAD) to Assess Effects on Vagal Tone and Strain Pressures Achieved Compared to a Standard Manometer in Healthy Volunteers Performing Standard and Modified Valsalva Manoeuvres.
Brief Title: Testing of a Valsalva Assist Device (VAD) in Healthy Volunteers Performing a Valsalva Manoeuvre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 1617/043
Record Dates: First submitted 2017-09-08; First posted 2017-10-02 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: SVT; Vagal Bradycardia
Keywords: Valsalva manoeuvre; Vagal tone; Modified Valsalva; Valsalva Assist Device
MeSH Terms: interventions — Supine Position; Patient Positioning

STUDY DESIGN:
Intervention Model Description: Four repeated measures in each participant in random order
Masking Description: Participants will not be able see manometer when using VAD Analysis of ECG traces will be blind to intervention as traces will be marked with a code, interventions carried out in random order and analysed in batches
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Four VM's (Other): Healthy volunteers undergo repeated VM's - Device: Supine VM VAD, Supine VAD manometer Modified VM VAD, Modified VM Manonmeter
  Interventions: Device: Supine VM VAD; Device: Supine VAD manometer; Other: Modified VM VAD; Other: Modified VM Manonmeter

INTERVENTIONS:
Device: Supine VM VAD — Valsalva strain delivered using VAD
  Other Names: Valsalva Assist Device supine
Device: Supine VAD manometer — supine Valsalva strain delivered using manometer
  Other Names: Valsalva Assist Device
Other: Modified VM VAD — modified VM using VAD
  Other Names: Standard (supine) position
Other: Modified VM Manonmeter — Postural modified position VM using manometer
  Other Names: Modified VM position

SUMMARY:
A prototype for a Valsalva Assist Device (VAD), which provides resistance to exhalation, has been developed and is ready for testing in healthy volunteers. There is a need to ensure the device can deliver the required strain and evaluate the physiological response (lowered heart rate) when used to deliver a Valsalva manoeuvre (VM) with and without postural modification.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the performance of a novel Valsalva assist device (VAD) in healthy volunteer and to confirm the physiological effects of a modified VM.

Specific Objectives:

To measure and compare peak strain pressure and duration produced using the device compared to a standard manometer in supine and modified postures

To evaluate whether there is a difference in vagal tone (drop in heart rate) in healthy volunteers performing a VM using the VAD versus manometer.

To evaluate whether there is a difference in vagal tone (drop in heart rate) in healthy volunteers performing a modified VM versus a standard supine VM using the VAD.

To evaluate whether there is a difference in vagal tone (drop in heart rate) in healthy volunteers performing a modified VM versus a standard supine VM using a manometer.

The investigators will conduct a single centre repeated measures observational study of use of the device to generate a Valsalva strain in a sample of healthy adult volunteers from the University of Exeter or RD&E Hospital staff. All participants will be screened for eligibility and undergo informed written consent prior to participation. If participants fail screening due to abnormal clinical readings or vital signs, the chief investigator will review them, any urgent abnormalities (very unlikely) would be reviewed by the chief investigator or delegated emergency department doctor as soon as they are discovered. Depending on the severity, if treatment is required urgently then they will be treated in the emergency department. Otherwise, they will be referred back to their GP. Potential participants will be given written information about the study at least 24 hours prior to recruitment and interested individuals invited to attend screening, recruitment and testing.

Potential participants will be invited to express an interest in taking part by responding to the trial poster. These posters will be displayed in the medical student common rooms ED department notice board. The potential participant contacts the researcher leading the practical aspects of the trial by phone or email. Respondents will be asked how they would like to receive further information (post, email, and phone) and offered an appointment at the Clinical Research Facility (CRF) for screening and written consent if eligible, at their convenience but at least 24 hours after receiving the information sheet. Given the simple, safe and quick nature of the interventions, participants will be given the choice to take part after written consent or to return on another date, whichever they would prefer, to ensure minimal visits whilst giving participants further time to consider taking part should they wish.

The VM is an extremely safe, physiological manoeuvre which is used in everyday life (eg straining at stool) and has been used in trial conditions and clinical practice many thousands of times with no serious adverse events. The investigators will exclude participants who could conceivably be at any risk of harm from performing a VM or from the use of the device.

The screening will include 12 lead ECG and physical examination including observations of heart rate, oxygen saturations, respiratory rate and blood pressure. Any participants with any detected abnormalities, whether they are excluded from participation or not, will be informed and referred to their primary care physician as appropriate. All testing will be conducted in the clinical research facility (CRF) of the Royal Devon & Exeter Hospital, according to a strict trial protocol.

Test Valsalva Manoeuvres:

Participants will undergo a total of 4 VMs of the following 4 variations in random order, stratified by method of strain generation to ensure balance between the order of manometer and device use:

1. Supine VM using a manometer. Supine Valsalva strain using a manometer visible to the participant with a target of 40mmHg for 15 seconds
2. Supine VM using the device. Supine Valsalva strain using the device connected to manometer invisible to the participant but visible to a researcher for 15 seconds
3. Modified VM using a manometer. Semi-recumbent (at 45 degrees) Valsalva stain using a manometer visible to the participant with a target of 40mmHg for 15 seconds followed by supine positioning and passive 45-degree leg lift immediately at the end of the strain for a further 15 seconds (the modified VM)
4. Modified VM using the device. Semi-recumbent (at 45 degrees) Valsalva strain using the device connected to manometer invisible to the participant but visible to a researcher for 15 seconds followed by supine positioning and passive 45-degree leg lift immediately at the end of the strain for a further 15 seconds (the modified VM)

ELIGIBILITY:
Inclusion Criteria:

* Adult Volunteers between 18 and 60 years old from University of Exeter or RD&E Hospital staff
* Sinus rhythm on initial ECG
* Self-reported good health

Exclusion Criteria:

* Any regular medication other than the oral contraceptive
* Previous cardiovascular or respiratory disease
* Any contraindication to performing a VM strain. (Eg. Known aortic stenosis, recent myocardial infarction, glaucoma, retinopathy)
* Pregnancy
* Any ECG abnormality
* Any contra-indication to postural modification (any reason the participant can't lie flat and have both legs lifted to 45 degrees, eg prosthetic hip
* Inability or refusal to give written consent to take part
* Observations of heart rate, oxygen saturations, respiratory rate or blood pressure outside the normal range. Specifically blood pressure less than 100 systolic
* Caffeinated drinks within 6 hours prior to testing
* The use of stimulant drugs or alcohol within 24 hours prior to testing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Appelboam, MBBS, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon & Exeter NHS FT, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] FitzGerald I, Ewings P, Lang I, Appelboam A. Testing of a novel Valsalva Assist Device with supine and modified positions in healthy volunteers. Emerg Med J. 2019 Jan;36(1):27-31. doi: 10.1136/emermed-2018-208004. Epub 2018 Dec 1. PMID 30504456

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Four VM's
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Four VM's
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 26.19 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 75

OUTCOME MEASURES:

1. Primary Outcome: Assessing Heart Rate During the Supine and Modified VM and Assessing Heart Rate While Using the VAD and Manometer
Description: Assessing the effects on heart rate of a supine valsalva manoeuvre compared to the modified Valsalva manoeuvres in healthy volunteers.The investigators will measure the longest RR (length between each r wave) length in mm during the 15 seconds during the manoeuvre and the 15 seconds afterwards on an 3 lead ECG trace. The investigators will measure pre strain heart rate using the 15 seconds of baseline heart rate before the maneouvre on the 3 lead ECG. Using an average of the RR length(mm). The heart rate in beats per minute will then be worked out using a calculation from the RR length. RR length (mm) x0.04 = RR in seconds. (10/RR in seconds)x60 = beats per minute. These arms are combined so as to make the data easier to understand. The higher the number the better the outcome. maximum score is minimum score is 25.9 with maximum 33.6
Time Frame: 3 minutes (4 repetitions of 45 seconds)
Measure: Mean (Full Range); unit: beat per minute
Groups:
- Mean Drop in Heart Rate Using the Modified VM: This measures the mean drop in heart rate before and after the modified valsalva manoeuvre using both the VAD and monometer
- Mean Drop in Heart Rate of Supine VM: This measures the mean drop in heart rate before and after the supine valsalva manouevre using the both the VAD and monometer
- Mean Drop in Heart Rate Using VAD: This measures the mean drop in heart rate before and after healthy participants undertook the modified and supine Valsalva manoeuvres while using the VAD
- Mean Drop in Heart Rate From Using the Manometer: This measures the mean drop in heart rate before and after healthy participants undertook the modified and supine Valsalva manoeuvres while using the manometer
Arm/Group | Mean Drop in Heart Rate Using the Modified VM | Mean Drop in Heart Rate of Supine VM | Mean Drop in Heart Rate Using VAD | Mean Drop in Heart Rate From Using the Manometer
Number analyzed (Participants) | 75 | 75 | 75 | 75
beat per minute | 33.6 [6.3 to 70.2] | 25.9 [5.4 to 61.2] | 28.7 [8.2 to 70.2] | 30.8 [5.4 to 61.2]
Statistical Analysis 1: Comparison: Mean Drop in Heart Rate Using the Modified VM vs Mean Drop in Heart Rate of Supine VM; Test type: Superiority; p < 0.001, mixed linear regression; Mean Difference (Net) = 3.7, 95% CI 2-sided [2.1 to 5.3], Standard Error of Mean 1.12
Statistical Analysis 2: Comparison: Mean Drop in Heart Rate Using the Modified VM vs Mean Drop in Heart Rate of Supine VM; Test type: Superiority; p = 0.003, mixed linear regression; Mean Difference (Net) = 2.3, 95% CI 2-sided [0.8 to 3.8]

2. Secondary Outcome: Percentage of Participants Who Acheived a 15 Second Strain Duration During a VM Comparing a Valsalva Assist Device and a Standard Manometer
Description: The investigators measured the time each Valsalva manoeuvre managed to keep to a 15-second drain if they managed 15 seconds at a pressure of 35-45mmHg this would count as an achieved strain.
Time Frame: 1 minute (4 repetitions of 15 seconds)
Measure: Count of Participants; unit: Participants
Groups:
- % Who Achieved 15 Second Strain Using a VAD: percentage of participants utilising the Valsalva assist device to achieve a valsalva manoeuvre who achieved the full 15 second strain using the Valsalva assist device
- % Who Achieved 15 Second Strain Using a Manometer: percentage of participants utilising the manometer to achieve a valsalva manoeuvre who achieved the full 15 second strain using the manometer
Arm/Group | % Who Achieved 15 Second Strain Using a VAD | % Who Achieved 15 Second Strain Using a Manometer
Number analyzed (Participants) | 75 | 75
Participants | 56 | 73

3. Secondary Outcome: Peak Sustained Pressure Testing of a Valsalva Assist Device (VAD) Compared to the Standard Manometer
Description: The investigators will measure the highest pressure achieved for more than a second using a manometer in mmHg and compare these done with the VAD and the manometer
Time Frame: 15 seconds (4 repetitions of 15 seconds)
Measure: Mean (Full Range); unit: mean (mmHg) of peak pressures acheived
Groups:
- Peak Pressures Acheived by VAD: peak pressure acheived by VAD
- Peak Pressures Acheived by Manometer: Peak pressures achieved by manometer
Arm/Group | Peak Pressures Acheived by VAD | Peak Pressures Acheived by Manometer
Number analyzed (Participants) | 75 | 75
mean (mmHg) of peak pressures acheived | 42.46 [30 to 50] | 39.96 [25 to 50]

ADVERSE EVENTS:
Time Frame: 15 minutes as each patient was taking part
Description: this was a very low risk study
Arm/Group | Four VM's
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 17/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Four VM's (N=75)
headache (Nervous system disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT03298880/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03298880/ICF_001.pdf